CLINICAL TRIAL: NCT02830048
Title: Low-dose Glibenclamide in Type 2 Diabetes Mellitus - Part A
Brief Title: Low dosE GlibENclamide in Diabetes Part A
Acronym: LEGEND-A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19062015; 2015-002837-23 (EudraCT Number)
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; glibenclamide; glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glibenclamide dose titration (Experimental): Increasing doses of glibenclamide oral suspension from 0.3mg/day to 6mg/day.
  Interventions: Drug: Glibenclamide

INTERVENTIONS:
Drug: Glibenclamide
  Other Names: GlibenTek

SUMMARY:
Diabetes is a chronic condition that affects 1 in 16 people in the UK, and leads to difficulty controlling blood sugar levels. This is due to an imbalance between two main hormones: insulin, which lowers blood sugar, and glucagon, which causes it to rise. Most current anti-diabetic medications work to improve insulin levels, however research is now shifting to better understand how glucagon levels play a key role in this disease.

Glibenclamide is a type of anti-diabetic medication (sulfonylurea) which is commonly used to increase the amount of insulin released by the pancreatic beta-cells. Studies in mice and human cells from donors with type 2 diabetes have shown that sulfonylureas can also improve glucagon levels when used in very small doses by working on different cells in the pancreas (alpha-cells).

The aim of this study is to find out whether low doses of glibenclamide can improve glucagon levels in patients with type 2 diabetes, and whether in the future this could be used to better control high blood sugar levels, without the risk of causing low blood sugar.

Participants with type 2 diabetes who are diet-controlled or on metformin will be given a liquid containing a low dose of glibenclamide. They will need to attend the OCDEM Clinical Research Unit at the Churchill Hospital, Oxford, for early morning blood tests every 3-4 days over a period of 3 weeks. A continuous glucose monitor will also be fitted during this time.

This study is funded by the NIHR OxBRC.

DETAILED DESCRIPTION:
This investigator-initiated clinical trial is a single-centre, open-label, non-randomised, dose-finding study. The am is to investigate whether treatment with low-dose glibenclamide can lead to a decrease in fasting glucagon levels in patients with type 2 diabetes, and whether this has an impact on overall blood glucose control.

It will be conducted in the Clinical Research Unit (CRU) of the Oxford Centre for Diabetes, Endocrinology and Metabolism (OCDEM) at the Churchill Hospital, Oxford. The aim is to find the dose of glibenclamide that causes a reduction in fasting glucagon levels in patients with T2DM.

Participants will self-administer increasing doses of an oral glibenclamide suspension from 0.3-6mg every 3 or 4 days, over a period of 21 days. They will attend the CRU for fasting pre-dose blood tests for insulin, glucagon, C- peptide and glucose prior to each dose change.

Additionally, participants will have the option of having a continuous glucose monitoring (CGM) sensor attached for the duration of the study, which will be checked and changed at each visit to CRU. This will measure the impact of treatment on overall blood glucose control.

No human trials have used doses of glibenclamide under 5mg previously in the measurement of insulin and glucagon secretion. Our sample size calculations are based on experimental data from isolated human islets from T2DM donors, which were performed in Professor Patrik Rorsman's lab. These suggest that 15 participants (allowing for a 15% dropout) would give the study 80% power to detect a 57% reduction in baseline glucagon levels with an alpha error of 5%.

Details of the study visits are as follows:

CRU visit 1 (1 hour):

1. Informed consent will be obtained by a member of the clinical trial team.
2. Inclusion and exclusion criteria checked.
3. Concomitant medication checked.
4. Demographics documented in case report form (CRF): date of birth, gender, weight, height.
5. Observations documented in CRF: resting heart rate and blood pressure.
6. Blood sample for HbA1c and safety blood tests (full blood count, renal function tests, electrolytes and liver function tests).
7. Pregnancy test in women of childbearing age (18-49 years old).
8. Participant informed to fast on next CRU visit.

CRU visit 2 (1 hour):

1. Observations documented in CRF: resting heart rate and blood pressure
2. Fasting blood sample for insulin, glucagon, C-peptide and glucose.
3. CGM sensor inserted.
4. Participants issued with oral glibenclamide suspension (0.6mg/ml) and dosing syringe. Educated on self-administration and given dosing schedule.

CRU visit 3 (30 minutes):

1. Observations documented in CRF: resting heart rate and blood pressure
2. Fasting blood sample for insulin, glucagon, C-peptide and glucose.
3. CGM sensor changed and data downloaded.

CRU visit 4 - 8 (30 minutes):

1. Observations documented in CRF: resting heart rate and blood pressure
2. Fasting pre-dose blood sample for insulin, glucagon, C-peptide and glucose.
3. CGM sensor changed and data downloaded.
4. Adverse event recording.
5. Check compliance. (visit 7 only: Participants issues with 6mg/ml oral glibenclamide suspension)

CRU visit 9 (30 minutes):

1. Observations documented in CRF: resting heart rate and blood pressure
2. Fasting pre-dose blood sample for insulin, glucagon, C-peptide and glucose.
3. CGM sensor removed and data downloaded. CGM system returned to CRU.
4. Adverse event recording.
5. Check compliance.
6. Unused oral glibenclamide suspension returned & document drug accountability.
7. Participants informed about end of study.

Telephone follow-up (15min):

Documentation of any adverse events occurred following the discontinuation of the trial medication.

Home visits:

For those participants not using the CGM and who are unable to attend the CRU for fasting blood tests, early morning home visits will be arranged. These will be conducted by a member of the research team and will replace CRU visits 3-9.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM.
* Age 18 years or over.
* Diet controlled or on metformin only for diabetic control.
* Body mass index 40 kg/m2 or less.
* HbA1c 6.0% to 9.5% (42mmol/mol to 80mmol/mol) inclusive.

Exclusion Criteria:

* Taking anti-diabetic therapies other than metformin
* Pregnancy or women of childbearing age without adequate contraception
* Women who are breastfeeding
* Major psychiatric disease including diagnosed eating disorders, history of drug or alcohol abuse
* Known sight-threatening retinopathy
* Renal impairment (eGFR < 60 ml/min; CKD Stage 3)
* Abnormal liver function tests (> 1.5 x upper limit of normal range)
* Known ischaemic heart disease or heart failure
* Known history of a stroke
* Known history of porphyria
* Concomitant use of miconazole or other oral antifungal medication.
* Known or suspected allergy to trial product or related products
* Oral steroid treatment 30 days prior to the start or at any time during the trial period.
* Known malignancy or any other condition or circumstance which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol.
* Ketoacidosis
* Felt to be unsuitable to participate in the trial in the opinion of the Chief Investigator.
* Receipt of any investigational trial drug within 3 month prior to participation in the current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Decrease in fasting plasma glucagon concentration | After 3-4 days of treatment at each dose increment
  Concentration of plasma glucagon using fasting blood samples prior to each dose change.

SECONDARY OUTCOMES:
Overall improvement in glycaemic control throughout the day | After 3-4 days of treatment at each dose increment
  Change in the percentage of Continuous Glucose Monitoring (CGM) readings under 4 mmol/L, between 4-10 mmol/L and above 10 mmol/L before starting glibenclamide and prior to each change in dose.
Effect on fasting glucose, insulin and C-peptide levels | After 3-4 days of treatment at each dose increment
  Concentration of glucose, insulin and C-peptide using fasting blood samples prior to each dose change.
Pre-dose plasma concentration of glibenclamide | After 3-4 days of treatment at each dose increment
  Concentration of plasma glibenclamide using fasting blood samples prior to each dose change.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Spiliotis, MD, Principal Investigator — University of Oxford
Locations (1):
- Clinical Research Unit, OCDEM, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The anonymised data (i.e. with studyID only) generated from this study will be deposited in the Oxford Research Archive (http://ora.ox.ac.uk/). This will provide a link between the results presented in publications and the underlying data. At the end of the retention period (currently 5 years), the data will be deleted from the archive.

REFERENCES:
- [Derived] Spiliotis II, Chalk R, Gough S, Rorsman P. Reducing hyperglucagonaemia in type 2 diabetes using low-dose glibenclamide: Results of the LEGEND-A pilot study. Diabetes Obes Metab. 2022 Aug;24(8):1671-1675. doi: 10.1111/dom.14740. Epub 2022 May 18. No abstract available. PMID 35491519